CLINICAL TRIAL: NCT03221166
Title: Thalidomide, a Novel Immunological Treatment to Modify the Natural History of Paediatric Crohn's Disease: a New Proposal From a Well-established Paediatric Research Network
Brief Title: Thalidomide Versus Infliximab in New Onset Crohn's Disease With Poor Prognostic Factors
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty in recruiting subjects who meet the inclusion/exclusion criteria
Sponsor: IRCCS Burlo Garofolo (Other)
Collaborators: Centro di Riferimento Oncologico - Aviano (Other); Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NET-2013-02355002
Record Dates: First submitted 2017-07-05; First posted 2017-07-18 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Crohn Disease
Keywords: Children; Crohn disease; Thalidomide; Mucosal healing
MeSH Terms: conditions — Crohn Disease | interventions — Thalidomide; Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thalidomide (Experimental): Thalidomide is a immunomodulatory and antiangiogenetic drug with anti tumor necrosis factor (TNF) alpha properties
  Interventions: Drug: Thalidomide
- Infliximab (Active Comparator): Infliximab is a chimeric monoclonal antibody against TNF alpha
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Thalidomide — Thalidomide is a immunomodulatory and antiangiogenetic drug with anti TNF alpha properties
  Arms: Thalidomide
Drug: Infliximab — Infliximab is a chimeric monoclonal antibody against TNF alpha
  Arms: Infliximab

SUMMARY:
Crohn's disease (CD) is a life-long inflammatory bowel disease disease with an unknown pathogenesis. The ultimate goal of therapy is to modify the natural history of CD thus reducing complications. Thalidomide is a small molecule with immunomodulatory and anti-angiogenetic properties. It is currently approved for the treatment of erythema nodosum leprosum, an immunological complication of leprosy and multiple myeloma. It has also been used in several other inflammatory diseases of the skin and of the mucosal membranes, such as Behcet disease, oropharyngeal ulcers in AIDS, cutaneous lupus, and graft versus host disease. Many case series and one pediatric randomized controlled trial proved the efficacy of thalidomide in the treatment of children with CD refractory to standard treatments. In these patients, clinical remission was achieved in about 50% of the cases and was maintained for a mean time superior of 3 years. Mucosal healing after 52 weeks of treatment was observed in 40% of the patients in clinical remission. Moreover, thalidomide was found to have a steroid-sparing effect and to decrease the need for surgical interventions. The clinical and endoscopic efficacy of thalidomide was also observed in children with failure to respond or intolerance to anti-TNF biological drugs.

The aim of this multicentric prospective randomized controlled is to evaluate the efficacy and safety of thalidomide vs infliximab in changing the natural history of CD in patients with poor prognostic outcome. Moreover, the study will evaluate the immunological and genetical mechanisms of CD, the mechanisms of action thalidomide in CD and will the pharmacokinetics, metabolomics and pharmacogenomics of thalidomide, and their impact on thalidomide safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age at diagnosis <18 years and >=6 years
* New diagnosis of CD based on Porto criteria
* CD with inflammatory phenotype (non-penetrating, non-fistulizing) and with no need for surgery except for perinal fistulas
* Presence of at least one of the following risk factors for poor prognosis:

  * fistulizing perianal disease
  * pan-enteric disease
  * disease extension > 60 cm
  * severe growth delay (height z-score < -2 DS)
  * severe osteoporosis (z score < -2 DS)
  * hypoalbuminemia (< 3g/dL) or high C-reactive protein (2 times higher the normal range)
* Acceptance of the Risk Evaluation and Mitigation Strategy (REMS) program for reducing the teratogenic risk.

Exclusion Criteria:

* ongoing pregnancy
* presence of peripheral neuropathy
* HIV
* patients with transplanted organs
* ongoing major infections or other severe diseases
* participation to other experimental studies.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Efficacy in inducing mucosal healing | 52 weeks
  Proportion of patients that achieve mucosal healing, defined by a Simplified Endoscopic Activity Index for CD (SES-CD) ≤ 2.

SECONDARY OUTCOMES:
Efficacy in inducing clinical response | 12 weeks
  Clinical response will be evaluated with the weighted Pediatric Crohn's Disease Activity Index (wPCDAI), defined by a reduction of wPCDAI > 50% from the basal values.
Efficacy in inducing clinical response | 52 weeks
  Clinical response will be evaluated with the weighted Pediatric Crohn's Disease Activity Index (wPCDAI), defined by a reduction of wPCDAI > 50% from the basal values.
Efficacy in inducing clinical remission | 12 weeks
  Clinical remission will be evaluated with the weighted Pediatric Crohn's Disease Activity Index (wPCDAI), defined by a wPCDAI <12.5.
Efficacy in inducing clinical remission | 52 weeks
  Clinical remission will be evaluated with the weighted Pediatric Crohn's Disease Activity Index (wPCDAI), defined by a wPCDAI <12.5.
Efficacy in reducing the need to change therapy | 12 weeks
  Evaluation of the proportion of patients that need a therapeutic change
Efficacy in reducing the need to change therapy | 52 weeks
  Evaluation of the proportion of patients that need a therapeutic change
Efficacy in reducing hospitalizations | 52 weeks
  Evaluation of the proportion of patients that need hospitalization.
Efficacy in reducing the need for surgery | 52 weeks
  Evaluation of the proportion of patients that need surgery
Efficacy in reducing erythrocyte sedimentation rate | Each time point between enrolment and 52 weeks (0, 4, 8, 14, 26, 38, 52 weeks)
  Evaluation of the trend of erythrocyte sedimentation rate (ESR)
Efficacy in reducing C-reactive protein | Each time point between enrolment and 52 weeks (0, 4, 8, 14, 26, 38, 52 weeks)
  Evaluation of the trend of C-reactive protein (CRP)
Efficacy in reducing faecal calprotectin | Each time point between enrolment and 52 weeks (0, 4, 8, 14, 26, 38, 52 weeks)
  Evaluation of the trend of faecal calprotectin
Efficacy in modifying body mass index | Each time point between enrolment and 52 weeks (0, 4, 8, 14, 26, 38, 52 weeks)
  Evaluation of the trend of body mass index, defined as weight (kg)/height (m)^2
Efficacy in modifying height-for-age z score | Each time point between enrolment and 52 weeks (0, 4, 8, 14, 26, 38, 52 weeks)
  Evaluation of the trend of height-for-age z score
Efficacy in modifying weight-for-age z score | Each time point between enrolment and 52 weeks (0, 4, 8, 14, 26, 38, 52 weeks)
  Evaluation of the trend of weight-for-age z score
Evaluation of the Treatment-Emergent Adverse Events | Between enrolment and 52 weeks
  Number and type
Direct and indirect costs | 52 weeks
  Comparison of direct and indirect costs (i.e. drugs, medical supplies and equipment, laboratory and diagnostic tests, hospitalizations, visits, transportation to and from healthcare facilities, missing work and school days…) between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Ventura, MD PhD, Study Chair — IRCCS Burlo Garofolo
Locations (6):
- Italy (6):
  - Dipartimento di Pediatria dell'Università di Napoli "Federico II", Napoli, Campania
  - IRCCS Burlo Garofolo, Trieste, Friuli Venezia Giulia
  - Pediatria III Gastroenterologia ed Endoscopia Digestiva, Istituto Giannina Gaslini, Genoa, Liguria
  - Fondazione MBBM , Azienda Ospedaliera San Gerardo - Università Milano Bicocca, Monza, Lombardy
  - Unità di Gastroenterologia Pediatrica e Fibrosi Cistica, Dipartimento di Scienze Pediatriche Mediche e Chirurgiche, Policlinico Universitario, Messina, Sicily
  - Gastroenterologia e Nutrizione Pediatrica, Azienda Ospedaliero Universitaria Meyer, Florence, Tuscany

IPD SHARING:
Plan to Share IPD: No